CLINICAL TRIAL: NCT03465969
Title: A Bioanalytical Method Cross-validation Study to Compare the Finger Prick Whole Blood MITRA Assay Method With the Established Venepuncture Whole Blood Method for Quantitative Determination of Tacrolimus Blood Concentrations in Transplant Patients
Brief Title: A Study to Compare the Finger Prick Whole Blood MITRA Assay Method With the Established Venepuncture Whole Blood Method for Quantitative Determination of Tacrolimus Blood Concentrations in Transplant Patients
Acronym: MITRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 506-MA-3189; 2017-004121-33 (EudraCT Number)
Record Dates: First submitted 2018-02-21; First posted 2018-03-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Kidney Transplantation; Liver Transplantation
Keywords: Kidney transplantation; A Bioanalytical Method Cross-validation; Advagraf; Liver transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver or kidney transplant participants of Advagraf (Other): Transplant participants will provide 1 whole blood venepuncture sample and 1 whole blood finger prick MITRA sample at pre-dose of participant's usual oral dose of commercial Advagraf and at approximately 1 and 3 hours post-dose.
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — oral
  Other Names: Advagraf

SUMMARY:
The purpose of this study is to assess relationship between tacrolimus concentrations determined via whole blood MITRA assay method with those determined using the established and validated whole blood venepuncture method using samples taken from liver and kidney transplant participants.

DETAILED DESCRIPTION:
This will be a bioanalytical assay method cross-validation study using blood samples donated by liver or kidney transplant participants. Participants will have been on a stable dose of Advagraf and deemed clinically stable for a period of 3-6 months and attend a routine out-patient follow-up visit to receive their usual oral dose of commercial Advagraf. Participants will be asked to provide 1 whole blood venepuncture sample and 1 whole blood finger prick MITRA sample at pre-dose and at approximately 1 and 3 hours post-dose. Participants will be kept at the study site for an extra 1 hour to ensure post-sampling safety and will be discharged thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subject will be a recipient of either a liver or kidney transplant and on a stable dose of commercial Advagraf minimum of 3 months.
* Subjects will be with clinically stable graft function for at least 3 months.

Exclusion Criteria:

* Subjects who are still participating in another clinical study or who have participated in a clinical study involving administration of an investigational drug in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Comparison of blood concentrations of tacrolimus | Day 1
  Tacrolimus concentrations will be determined from the dried whole blood samples collected via finger prick into MITRA cartridge and in whole blood taken by venipuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Physician, Study Director — Astellas Pharma Europe Ltd.
Locations (4):
- France (2):
  - Site FR33002, Toulouse
  - Site FR33001, Villejuif
- United Kingdom (2):
  - Site UK44002, Cambridge
  - Site UK44001, London

IPD SHARING:
Plan to Share IPD: Undecided